CLINICAL TRIAL: NCT03989050
Title: Immunogenicity and Safety of Pneumococcal Vaccination in Patients Treated With Immune Checkpoint Inhibitors
Acronym: SPICE
Status: Withdrawn | Type: Observational
Why Stopped: Administrative reasons
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Sibylle C Mellinghoff, Dr. med., University of Cologne
Other Study IDs: SPICE
Record Dates: First submitted 2019-06-13; First posted 2019-06-18 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Melanoma; Non Small Cell Lung Cancer
Keywords: Immune Checkpoint Inhibitor; Pneumococcal Vaccination
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be obtained for determination of pneumococcal antibody-titers during clinical routine care. One sample will be drawn before vaccination. After 30 days, a second blood sample will be taken during an already planned visit at the (outpatient) clinic. Titer assessment will be performed along STIKO recommendations for immunocompromised patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Melanoma patients: Patients receiving therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) agent for melanoma
- Non-small cell lung cancer (NSCLC) patients: Patients receiving therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) agent for NSCLC
- other malignancy patients: Patients receiving therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) agent for other malignancy

SUMMARY:
This is a prospective observational study of vaccine efficacy and safety in adult patients with malignancies (melanoma/Hodgkin's lymphoma/Non-small cell lung cancer). The primary objective is to compare serotype specific immunoglobulin G (IgG) antibody titres before and after pneumococcal vaccination in patients receiving Immune Checkpoint Inhibitors (ICI). As an explorative objective, serotype specific IgG antibodies measured by ELISA and those measured by Opsonophagocytosis assay (OPA) after pneumococcal vaccination in patients receiving ICI will be correlated. In addition, the incidence of immune related adverse events (irAE) in patients vaccinated during ICI treatment will be determined.

DETAILED DESCRIPTION:
Physicians will be informed by mail and pocket cards with all necessary information about the study, in particular eligibility criteria. Patients currently receiving Immune Checkpoint Inhibitors will be approached by their treating physicians in case of an already scheduled vaccination against S. pneumonia. If a patient agrees to participate in the study and to sign an informed consent form, basic data on demographics, underlying disease, comorbidities, and irAE will be obtained from the electronic health record and entered into the eCRF.

Pneumococcal antibody titers will be drawn at baseline and after 30 days. We will actively follow-up on study patients for four months after enrolment and screen health records of the enrolled patients after four months to record occurrence of irAE.

A blood sample (9 ml) will be drawn before vaccination. Vaccination will either be performed by the treating physician or by a general practitioner. After 30 days, a second blood sample will be taken during an already planned visit at the (outpatient) clinic. Titer assessment will be performed along STIKO recommendations for immunocompromised patients.

All samples for ELISA and OPA titer determination will be stored frozen at Department I for Internal Medicine and titers will be analyzed in batch at the end of this study. All therapies and diagnostics including vaccinations will be administered solely as part of clinical routine and as recommended by appropriate guidelines (RKI STIKO recommendations).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age ≥18 years
* Receiving pneumococcal vaccination for the first time along STIKO criteria
* Therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) agentfor melanoma, NSCLC or other malignancy

Exclusion Criteria:

* Patients unwilling/ineligible for vaccination under current STIKO recommendations
* Previous vaccination with any licensed or experimental pneumococcal vaccine
* Concurrent treatment with anti-CTLA-4 agent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients treated with ICI (for melanoma, NSCLC, or other malignancy), vaccinated against S. pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Pneumococcal antibody kinetics | 1 Month
  Comparison of serotype specific IgG antibody titers before and after pneumococcal vaccination in patients receiving ICI

SECONDARY OUTCOMES:
Determination of applicability of current assessment methodology | 1 year
  Correlation of serotype specific IgG antibodies measured by ELISA and those measured by OPA after pneumococcal vaccination in patients receiving ICI
Incidence of irAE | 1 year
  Assessment of the incidence of irAE in patients vaccinated during ICI treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle C Mellinghoff, MD, Principal Investigator — University of Cologne
Locations (2):
- Germany (2):
  - University Hospital Cologne, Cologne, North Rhine-Westphalia
  - HELIOS University Hospital Wuppertal, Wuppertal, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: Undecided